CLINICAL TRIAL: NCT02290054
Title: Auriculotherapy for Prevention of Postoperative Urinary Retention in Men Receiving Postoperative Epidural Analgesia After Thoracic Surgery
Brief Title: Auriculotherapy for Prevention of Postoperative Urinary Retention
Acronym: RUPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013/41; 2013-A01396-39 (Other: ANSM)
Record Dates: First submitted 2014-11-08; First posted 2014-11-13 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Analgesia, Epidural
Keywords: analgesia, epidural; urinary retention
MeSH Terms: conditions — Agnosia; Urinary Retention | interventions — Therapeutics; Auriculotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): A thoracic epidural catheter is inserted first. Then total intra-venous anesthesia is performed. Implementation of adhesive pads on the ears is performed while the patient is sleeping but before thoracic incision.
  Interventions: Procedure: Control; Procedure: Intra-venous anesthesia
- Treated (Experimental): A thoracic epidural catheter is inserted first. Then total intra-venous anesthesia is performed. Auriculotherapy is performed while the patient is sleeping but before thoracic incision.
  Auriculotherapy uses semi-permanent needles and implementation of adhesive pads to mask the needles.
  Interventions: Procedure: Treated; Procedure: Intra-venous anesthesia

INTERVENTIONS:
Procedure: Control — Implementation of adhesive pads on the ears is performed while the patient is sleeping but before thoracic incision.
  Other Names: Sham Comparator
  Arms: Control
Procedure: Treated — Auriculotherapy uses semi-permanent needles and implementation of adhesive pads to mask the needles.
  Other Names: Auriculotherapy
  Arms: Treated
Procedure: Intra-venous anesthesia

SUMMARY:
Urinary retention is a common complication of epidural analgesia. Auriculotherapy could prevent this complication. This study will be performed among men receiving thoracic epidural analgesia after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to a lung surgical procedure and thoracic epidural analgesia

Exclusion Criteria:

* Abnormalities of the external ear
* Dialysis or end stage renal failure
* Abnormal urinary tract
* Incapacity to self assessment of comfort and anxiety,
* Contra-indication to total intravenous anesthesia

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

PRIMARY OUTCOMES:
bladder catheterization | 24 hours
  Requirement of bladder catheterization during the day and the first night following surgery

SECONDARY OUTCOMES:
Comfort | 24 hours
  The degree of patient's comfort is assessed six hours after his arrival in the recovery room and the morning after surgery using a numerical scale from 0 '"maximum discomfort " to 10" maximum comfort "
Anxiety | 24 hours
  The degree of patient's anxiety is assessed six hours after his arrival in the recovery room and the morning after surgery using a numerical scale from 0 '"maximum discomfort " to 10" maximum comfort "

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hôpital Foch, Suresnes, Hauts de Seine, France

REFERENCES:
- [Derived] Michel-Cherqui M, Szekely B, Lemoyne F, Feliot E, Gayat E, Fischler M. Auriculotherapy in the prevention of postoperative urinary retention in patients with thoracotomy and thoracic epidural analgesia: A randomized, double-blinded trial. Medicine (Baltimore). 2019 Jun;98(23):e15958. doi: 10.1097/MD.0000000000015958. PMID 31169723